CLINICAL TRIAL: NCT05925621
Title: Cognitive Neurology Unit's Anti-amyloid Monoclonal Antibodies for the Treatment of Alzheimer's Disease Clinical Registry
Brief Title: Cognitive Neurology Unit Clinical Registry
Status: Recruiting | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Daniel Press, Chief, Cognitive Neurology Unit, Beth Israel Deaconess Medical Center
Other Study IDs: 2023P000494
Record Dates: First submitted 2023-06-22; First posted 2023-06-29 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — lecanemab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Lecanemab: Patients with Alzheimer Disease receiving anti-amyloid mAb therapy at the BIDMC
  Interventions: Drug: Lecanemab

INTERVENTIONS:
Drug: Lecanemab — Observational study

SUMMARY:
A Prospective Comparative Study Of Monoclonal Antibodies For The Treatment Of Alzheimer's Disease

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is a neurodegenerative disorder associated with brain deposition of extracellular amyloid and intracellular tau. It causes progressive cognitive impairment, especially memory, and is invariably fatal. Currently, there is no effective treatment for AD. A new and promising method involves the use of anti-amyloid-beta monoclonal antibodies (anti-amyloid mAbs) to reduce amyloid accumulation in brain. There are currently two anti-amyloid mABs, aducanumab and lecanemab, approved by the FDA under FDA's "accelerated approval" pathway. However, so far there is only a single phase 3 study that unequivocally demonstrates clinical efficacy of anti-amyloid mAB therapy1. This study is designed to help determine the therapeutic benefit of anti-amyloid mABs therapy by treating AD patients in our clinic with anti-amyloid mABs and measuring cognitive impairment and functional outcomes over the course of the treatment period and beyond. This study has 4 specific aims.

SPECIFIC AIM 1: TO CREATE A CNU ANTI-AMYLOID MONOCLONAL ANTIBODY REGISTRY

SPECIFIC AIM 2: TO DETERMINE WHETHER ANTI-AMYLOID MABs SLOW COGNITIVE AND FUNCTIONAL DECLINE

SPECIFIC AIM 3: TO IDENTIFY ANY ASSOCIATIONS BETWEEN SIDES EFFECTS AND PATIENT CHARACTERISTICS

SPECIFIC AIM 4: TO ESTABLISH THE TIME COURSE OF CLINICAL BENEFITS

ELIGIBILITY:
Inclusion Criteria:

* o Patient meets clinical criteria for mild cognitive impairment or early dementia from Alzheimer's disease

  * Patient has evidence of cognitive impairment on neuropsychological testing
  * Patient has not progressed to the moderate stage of dementia based on neuropsychological testing or clinical judgement
  * Amyloid PET imaging and/or CSF analysis consistent with Alzheimer's disease
  * Amyloid PET imaging positive
  * CSF p-Tau/Abeta42 ration >0.023 and ABeta42 < 1027**
  * 3T MRI in past 6 months
  * Patient has a care partner
  * Patient under the care of an appropriate BI-Lahey amyloid clinic
  * Patient is on a stable medication regimen

Exclusion Criteria:

* o Recent stroke or suspected TIA in the past year

  * Pregnancy
  * Active autoimmune or immunological disease
  * Systemic treatment with immunosuppressants, immunoglobulins, or monoclonal antibodies or their derivatives
  * Bleeding disorder with Plts < 50,000 or INR > 1.5
  * On warfarin, heparin, or DOAC
  * On dual antiplatelet therapy
  * Non Alzheimer disease cause of dementia/MCI
  * ApoE e4 homozygote

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will enroll patients under the care of the CNU. All patients with a concern for cognitive impairment secondary to AD interested in receiving anti-amyloid monoclonal antibody therapy will be enrolled into this registry as required by CMS.
  * Patients with a diagnosis of AD based on National Institute on Aging and the Alzheimer's Association diagnostic guidelines.
  * Patients with a diagnosis of MCI based on the National Institute on Aging and the Alzheimer's Association and Petersen criteria.
  * All patients eligible to receive anti-amyloid therapy will have confirmation of AD through a positive amyloid PET.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-07-16 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
To Determine Whether Anti-Amyloid Mabs Slow Cognitive And Functional Decline | 30 months
  This study is a prospective, registry-based, single unit, observational study comparing clinical outcome in patients receiving anti-amyloid mAb therapy to historical norms.
To Identify Any Associations Between Side Effects And Patient Characteristics | 30 months
  This study is a prospective, registry-based, single unit, observational study comparing anti-amyloid mAb therapy patient demographics to clinical outcomes.
To Establish The Time Course Of Clinical Benefits | 30 months
  This study is a prospective, registry-based, single unit, observational study examining anti-amyloid mAb therapy patient clinical outcomes and adverse effects over time.

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sets may be shared with members outside the study team following de-identification under approved data use agreements (DUAs) as needed. Within the REDcap database, access to the identifiable information will be limited to study staff members and to staff managing the database. Any data that may require a physical transfer from one place to another will be done using removable encrypted data storage devices.
Supporting Information: CSR